CLINICAL TRIAL: NCT00456664
Title: Molecular Diagnostics for CMV Disease and IRIS in HIV-1 Infected Persons, and the Mechanism Study for CMV Alternative Gene Splicing in Immediate Early Protein
Brief Title: CMV Disease and IRIS in HIV-1 Infected Persons
Status: Completed | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Other Study IDs: QM094007
Record Dates: First submitted 2007-04-04; First posted 2007-04-05 (Estimated); Last update posted 2009-02-03 (Estimated); Status verified 2008-05

CONDITIONS: HIV Infections; Cytomegalovirus
Keywords: CMV; IRIS
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Genetic: IE gene

SUMMARY:
Various diagnostic methods are available for CMV infection. But none of them could be a standard and highly valuable. Our first goal is to setup a series of molecular diagnostic tools for HIV-1 infected person. By using these tools, physicians can easily select cases with CMV disease or immune restoration inflammatory syndrome (IRIS) to enroll this study. Furthermore, we will seek for a predict marker for CMV reactivation, CMV disease and IRIS. Finally, our research will focus on the mechanism of the IE gene alternative splicing between lytic and latent stage.

DETAILED DESCRIPTION:
At present, human cytomegalovirus (HCMV) remains a major health threat in immune compromised patients. Especially HCMV will cause blind and death in HIV-1 infected person. Currently, few antiviral drugs can be chosen for treatment of HCMV infection. Besides, more and more drug resistant virus strains were reported and led failure in antiviral therapy.

Various diagnostic methods are available for CMV infection. Such as shell vial assay, CMV antigen test, pp65 antigen assay and polymerase chain reaction. But none of them could be a standard and highly valuable. Although CMV-PCR is very sensitive, it can't distinguish between active disease and asymptomatic infection or latency, can't predict symptomatic disease nor can't monitor the successful antiviral therapy.

Our first goal is to setup a series of molecular diagnostic tools for HIV-1 infected person. By using these tools, physicians can easily select cases with CMV disease or immune restoration inflammatory syndrome (IRIS) to enroll this study. Furthermore, we will seek for a predict marker for CMV reactivation, CMV disease and IRIS. Finally, our research will focus on the mechanism of the IE gene alternative splicing between lytic and latent stage. We may find out new therapeutic concept and prevent virus reactivation from latency.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of HIV-1 Disease
* Clinical diagnosis of CMV disease or immune restoration inflammatory syndrome (IRIS)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2006-11; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jih-Jin Tsai, M.D., Study Director — Chung-Ho Memorial Hospital,Kaohsiung Medical University
Locations (1):
- Kaoshing Medical University Chung-Ho Memorial Hospital, Kaoshiung, Taiwan